CLINICAL TRIAL: NCT07083414
Title: Impact of Digital Oral Health Educational Program on a Group of Geriatrics Oral Health and Quality of Life Compared to Standard Oral Health Educational Program in Egypt: a Cluster Randomized Control Trial
Brief Title: Impact of Digital Oral Health Educational Program on a Group of Geriatrics Oral Health and Quality of Life Compared to Standard Oral Health Educational Program in Egypt
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Weam abdelhamid hassab elnaby elshoura, The principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Edu. Program
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Oral Health Self-efficacy; Healthy Participants Study
Keywords: Educational program; Oral health program; Quality of life

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elderly participant will receive digital educational oral health program. (Experimental): The digital oral health educational program will be through 6 months and follow up 3 times every 1.5 months through this period. The content will focus on age-related oral health changes, oral hygiene practices, denture care, and disease prevention.
  Interventions: Device: elderly participant will receive digital educational oral health program.
- elderly participant will receive the standard oral health education in geriatric institution. (Active Comparator): Participants in the control group will receive standard oral health information. No education sessions will be conducted during the 6 months till the final assessment. However, after the final assessment at 6 months, the control group will be offered access to the digital educational program.
  Interventions: Other: elderly participant will receive the standard oral health education in geriatric institution.

INTERVENTIONS:
Device: elderly participant will receive digital educational oral health program. — * Digital 3D Model Video: A custom-designed 3D animated video illustrating proper tooth brushing techniques tailored for elderly individuals, as well as comprehensive guidance on denture care.
  * Written Educational Materials: Printed resources including posters and flyers that provide key messages and visual demonstrations related to maintaining good oral hygiene practices.
  * PowerPoint Presentations and Educational Videos: Visual and audiovisual materials focusing on the importance of balanced nutrition in maintaining oral and general health, and early detection of oral cancer, including risk factors, signs, and recommended screening practices.
  * Hands-on Brushing Technique Training: Practical sessions utilizing dental cast models to demonstrate and allow participants to practice effective brushing techniques under supervision.
  Other Names: Digital oral health educational program
  Arms: elderly participant will receive digital educational oral health program.
Other: elderly participant will receive the standard oral health education in geriatric institution. — The use of traditional health promotion materials, such as leaflets and posters, remains valuable in community settings. These tools are cost-effective, easy to produce, and continue to serve as effective educational resources for adults, including the elderly. Participants in the control group will receive standard oral health information. No education sessions will be conducted during the 6 months till the final assessment. However, after the final assessment at 6 months, the control group will be offered access to the digital educational program.
  Other Names: Standard oral health educational program
  Arms: elderly participant will receive the standard oral health education in geriatric institution.

SUMMARY:
The aim of the study is to evaluate the impact of a digital oral health education program on the oral health status and quality of life for geriatric populations compared to standard oral health education in Egypt.

DETAILED DESCRIPTION:
The principal investigator will carry out all educational programs.

For both interventions:

* Informed consent from elderly participating.
* Baseline records plaque index(Appendix : silness and loe), WHO questionnaire (Appendix : oral health survey) and GOHAI (Appendix : Geriatric Oral Health Assessment Index).
* Allocation (The outcome will be immediately recorded and sealed in a numbered, opaque envelope corresponding to the cluster. These envelopes will only be opened after the cluster has been enrolled in the study, thus preventing any fore knowledge of the allocation and reducing the risk of selection bias).
* Examination will be performed to assess the inclusion criteria.

All geriatric institution will then be allocated into either one of the groups alternatively depending on the educational program used as follows:

Group I (Experimental group); elderly participant will receive digital educational oral health program.

Group II (Control group); elderly participant will receive the standard oral health education in geriatric institution.

. Group I (Experimental group); elderly participant will receive digital educational oral health program.

The digital oral health educational program will be through 6 months and follow up 3 times every 1.5 months through this period. The content will focus on age-related oral health changes, oral hygiene practices, denture care, and disease prevention.

Digital 3D model video designed for the elderly population. Posters Flyers Power-point Cast model Educational videos

. Group II (Control group); elderly participant will receive the standard oral health education in geriatric institution. Participants in the control group will receive standard oral health information. No education sessions will be conducted during the 6 months till the final assessment. However, after the final assessment at 6 months, the control group will be offered access to the digital educational program.

ELIGIBILITY:
Inclusion Criteria:

* Old age population above years old.
* Participants who is willing to confirm consent for the educational program and assessment.
* Participants without disability that interfere during communication.

Exclusion Criteria:

* Individuals with palliative care and rehabilitation ward, presence of mental disorder, had dangerous communicable disease.
* Participants who refused to participate.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Dental plaque | Assessed at baseline and after 6 months
  It measures the thickness of dental plaque at the gingival area by using dental mirror and pen light then score ranging from to per tooth surface.
  0= absence of microbial plaque
  1. thin film of microbial plaque along the free gingival margin
  2. moderate accumulation with plaque in sulcus
  3. large amount of plaque in sulcus or pocket along with free gingival margin

SECONDARY OUTCOMES:
General oral health status (WHO oral health assessment form for adult, 2013) | Assessed at baseline and after 6 months
  Use form to evaluate oral hygiene practices, dental needs, and clinical oral conditions. This tool assesses multiple oral health domains, including the condition of the dentition (such as decayed, filled, or missing teeth), periodontal status using the modified Community Periodontal Index (CPI), loss of attachment, dental erosion, dental trauma, enamel fluorosis, oral mucosal lesions, denture presence, and treatment urgency. For periodontal status (CPI), scores range from 0 to 4, where 0 indicates a healthy condition, and higher scores reflect increasing severity, such as bleeding, calculus presence, and periodontal pocket depth (up to 6 or more). Similarly, loss of attachment is scored from 0 to 4, with higher values indicating greater tissue destruction (ranging from 0-3 up to 12 mm). Other conditions such as erosion, trauma, and mucosal lesions are recorded based on presence or severity. Higher scores in the periodontal and attachment domains indicate worse oral health conditions.

OTHER OUTCOMES:
Oral health- related quality of life | Assessed at baseline and after 6 months
  Geriatric oral health assessment index (GOHAI) 12 items validated questionnaire in Arabic assessing the impact of oral health on physical function, psychosocial function, and pain/discomfort with (0-5)score as 0= minimum and better oral health quality of life and 5= maximum and worse oral health quality of life 0= never 1= rarely 2= sometimes 3= often 4= a lot 5= always

IPD SHARING:
Plan to Share IPD: No